CLINICAL TRIAL: NCT02928302
Title: Transvaginal Ultrasound Cervical Length Screening in Singleton Pregnancy Without Prior Spontaneous Preterm Birth
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: new protocol started 31/18
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, MD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 254/16
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TVU CL screening (Experimental): TVU CL screening: single TVU CL at 18 0/7 to 23 6/7 every week
  Interventions: Other: TVU CL screening
- no screening (No Intervention): no TVU CL screening

INTERVENTIONS:
Other: TVU CL screening — Transvaginal ultrasound cervical length screening
  Arms: TVU CL screening

SUMMARY:
Preterm birth (PTB) is a major cause of perinatal morbidity and mortality. Worldwide, about 15 million babies are born too soon every year, causing 1.1 million deaths, as well as short- and long-term disability in countless survivors. Few prognostic tests are available to predict PTB. A short transvaginal ultrasound cervical length (TVU CL) has been shown to be a good predictor of PTB.Different strategies have been adopted for prevention of PTB. The evidence supports the use of vaginal progesterone in singleton pregnancies with short cervix, while cervical cerclage seems to be beneficial only in the subgroup of singleton gestations with both prior spontaneous PTB and TVU CL ≤25mm, and not in singletons without prior PTB, nor in multiple gestations.

However, so far there are no level-1 data on the efficacy of TVU CL screening neither in low risk nor in high risk pregnancy Thus, we aim to assess the efficacy of a policy of TVU CL screening in singleton pregnancy without prior spontaneous PTB

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Singleton pregnancy (limits the participants to female gender)
* No prior spontaneous preterm delivery, defined as spontaneous preterm delivery 16 0/7 - 36 6/7 weeks

Exclusion Criteria:

* Multiple gestation
* Prior spontaneous preterm birth 16-36 6/7 weeks
* Ruptured membranes at time of randomization
* Lethal fetal structural anomaly at time of randomization
* Fetal chromosomal abnormality at time of randomization
* Placenta previa and/or accreta at time of randomization
* Women who already underwent TVU CL measurement during the index pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
preterm birth rate | Less than 37 weeks
  either spontaneous or indicated preterm delivery

SECONDARY OUTCOMES:
Perinatal death | Between birth and 28 days of age
  either neonatal death or fetal death
preterm birth rates | Less than 24, 28, 32, 30, and 34 weeks gestation
  either spontaneous or indicated preterm delivery
admission to neonatal intensive care unit | time of delivery
Composite perinatal outcome | Between birth and 28 days of age
  Includes necrotizing enterocolitis (NEC), intraventricular hemorrhage (IVH) (grade 3 or higher), respiratory distress syndrome (RDS), bronchopulmonary dysplasia (BPD), retinopathy (ROP), blood-culture proven sepsis and neonatal death
necrotizing enterocolitis | Between birth and 28 days of age
  Defined as modified Bell Stage 2 or 3. Stage 2: Clinical signs and symptoms with pneumatosis intestinalis on radiographs. Stage 3: Advanced clinical signs and symptoms, pneumatosis, impending or proven intestinal perforation
intraventricular hemorrhage (grade 3 or higher) | Between birth and 28 days of age
  IVH
respiratory distress syndrome | Time of delivery
  Respiratory distress with an oxygen requirement and a chest x-ray that shows hypoaeration and reticulogranular infiltrates
birth weight | time of delivery
Length of hospital stay | Discharge from hospital
  Days in NICU
Neonatal death | Between birth and 28 days of age
gestational age at delivery | time of delivery
latency | time of delivery
  from randomization to delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Saccone, Naples, Italy

IPD SHARING:
Plan to Share IPD: No